CLINICAL TRIAL: NCT03000465
Title: Individualized Pneumoperitoneum Pressure in Colorectal Laparoscopic Surgery Versus Standard Therapy (IPPCollapse-I)
Brief Title: Individualized Pneumoperitoneum Pressure in Colorectal Laparoscopic Surgery
Acronym: IPPCollapseI
Status: Completed | Type: Observational
Sponsor: Hospital Universitario La Fe (Other)
Collaborators: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Principal Investigator, Oscar Diaz-Cambronero, Physician, specialist in Anesthesiology, Hospital Universitario La Fe
Other Study IDs: 2015/0094
Record Dates: First submitted 2016-12-15; First posted 2016-12-22 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Individualized Pneumoperitoneum Pressure
Keywords: pneumoperitoneum pressure; laparoscopic pressure; intra-abdominal insufflation; intra-abdominal pressures; abdominal compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients undergoing laparoscopic colorectal surgery
  Interventions: Procedure: Laparoscopic colorectal surgery

INTERVENTIONS:
Procedure: Laparoscopic colorectal surgery — Minimizing intra-abdominal insufflation pressure in laparoscopic colorectal surgery as an individualized strategy

SUMMARY:
Optimizing all factors that increase the intra-abdominal volume and performing an individualized strategy should allow us to reduce the pneumoperitoneum insufflation pressure while maintaining optimal surgery conditions for a laparoscopic colorectal surgery, compared to the standard strategy of maintaining fixed intra-abdominal insufflation pressures (12-15 mmHg).

DETAILED DESCRIPTION:
In the context of multimodal rehabilitation in colorectal laparoscopic surgery (Fast Track or ERAS (Enhance Recovery After Surgery)) multiple strategies have been introduced that have managed to improve patient recovery, decrease postoperative complications, decrease hospital days and decrease the overall costs per process.

The possibility of performing individualized colorectal laparoscopic surgery with the minimum insufflation pressure guaranteeing optimal surgical conditions has not been evaluated and this would allow us to reduce the impact of surgery on the patient, decrease perioperative morbidity and improve patient recovery.

In our study, abdominal compliance, Pv0 and maximal Pv were determined during the initial performance of the pneumoperitoneum, and then a stepwise protocol for the reduction of intra-abdominal pressure (IAP) insufflation was stablished with evaluation by the surgeons, until reaching the minimal insufflation IAP in which optimal surgical conditions are maintained.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* ASA I-III (American Society of Anesthesiologists physical status classification)
* Signed informed consent
* Absence of cognitive deficit

Exclusion Criteria:

* Urgent surgery
* Pregnancy or breastfeeding
* Immune Disorder
* Advanced renal, hepatic or cardiopulmonary disease
* Negative to participate in the study
* Under 18 years
* Inability to give consent
* Associated neuromuscular disorders
* Allergy to rocuronium/sugammadex
* Contraindication for use of rocuronium/sugammadex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing colorectal laparoscopic surgery. Patients will be excluded of the analysis if the surgery cannot be finished by laparoscopy,
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2015-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Minimal intra-abdominal pressure | From pneumoperitoneum induction until surgery completion (during the intraoperative period), up to 300 minutes.
  To obtain values of intra-abdominal pressure level of minimum insufflation that guarantees optimal surgical conditions following an individualized strategy [mmHg].

SECONDARY OUTCOMES:
Ventilation pattern pressure | From pneumoperitoneum induction until surgery completion (during the intraoperative period), up to 300 minutes.
  Airway pressures at different levels of IAP (peak pressure, PEEP (positive end expiratory pressure), plateau pressure, driving pressure) [mmH2O].
Intra-abdominal pressures (Pv0, maximal IAP) | From pneumoperitoneum induction until surgery completion (during the intraoperative period), up to 300 minutes.
  Pv0 (IAP with volume 0) and maximal IAP [mmHg].
Intra-abdominal pressures (abdominal compliance). | From pneumoperitoneum induction until surgery completion (during the intraoperative period), up to 300 minutes.
  Dynamic abdominal compliance per liter (DV/DP, difference in volume/difference in pressure [L/mmHg]).
Surgeon skills and experience | Years of experience, up to 10 years.
  Previous experience of the surgeon in laparoscopic surgery, annual cases, years of experience, previous experience with low IAP.
Duration of surgery | The follow-up period will be extended during the intraoperative period, from initial incision until surgery completion, up to 300 minutes.
  Duration of surgery in minutes from incision to abdominal wall closure.
Postoperative complications | The follow-up period will be extended until hospital discharge for the evaluation of complications, an average of 7 to 10 days.
  Evolution and complications in the postoperative period: Postoperative pain in the first 24 hours. Postoperative complications were assessed using the Clavier-Dindo classification.
Hospital stay | The follow-up period will be extended until hospital discharge for the evaluation of complications, an average of 7 to 10 days.
  Hospital stay in days

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Diaz Cambronero, Principal Investigator — Physician, Specialist in Anesthesiology

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Diaz-Cambronero O, Flor Lorente B, Mazzinari G, Vila Montanes M, Garcia Gregorio N, Robles Hernandez D, Olmedilla Arnal LE, Argente Navarro MP, Schultz MJ, Errando CL; IPPColLapSe study group. A multifaceted individualized pneumoperitoneum strategy for laparoscopic colorectal surgery: a multicenter observational feasibility study. Surg Endosc. 2019 Jan;33(1):252-260. doi: 10.1007/s00464-018-6305-y. Epub 2018 Jun 27. PMID 29951750